CLINICAL TRIAL: NCT01612572
Title: A Registry Study on Safety Surveillance of Xiyanping (a Chinese Medicine Injection) Used in China
Brief Title: A Registry Study on Xiyanping(a Chinese Medicine Injection) Used in Fifty Hospitals
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yanming Xie, Deputy Director, China Academy of Chinese Medical Sciences
Other Study IDs: RSCMI-Ⅲ; RSCMI- Ⅲ
Record Dates: First submitted 2012-06-03; First posted 2012-06-06 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Viral Pneumonia; Bronchitis; Infantile Diarrhea; Bacillary Dysentery; Virus Hepatitis
MeSH Terms: conditions — Pneumonia, Viral; Bronchitis; Diarrhea, Infantile; Dysentery, Bacillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study was advocated by Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences in October 2011.

It was funded by China major scientific and technological specialized project for 'significant new formulation of new drugs'.

Xiyanping is kind of Chinese Medicine injection used for treating viral pneumonia 、bronchitis、amygdalitis、infantile diarrhea、bacillary dysentery 、virus hepatitis、and Children acute hot diseases in many Chinese hospitals.

The purpose of this study is to determine adverse drug events or adverse drug reaction in large sample size 20,000 patients.

DETAILED DESCRIPTION:
It is very common that Chinese Medicine Injection used in hospitals in mainland China. However safety problems rose in recent years. There could be many uncertain factors influence Chinese Medicine Injection in clinical practice.

In order to ensure the safety of public drug use and lower drug-induced risks, a registry study for Xiyanping injection safety surveillance with 20000 patients will be conducted from Jan.2012 to Dec.2015.

Eligibility criteria Patients who will use Xiyanping injection in selected hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Xiyanping injection from 2012 to 2014

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An anticipated sample size was caculated in this study, about 20000. Patients using Xiyanping injection from 2012 to 2014 in more than 50 hospitals
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events; incidence of Xiyanping'ADRs and identify factors that contributed to the occurrence of the adverse reaction | The registry procedure will last 3 years only for patients using Xiyanping.

CONTACTS AND LOCATIONS:
Overall Officials: Yan M Xie, BA, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences